CLINICAL TRIAL: NCT05914285
Title: Assessment of Salbutamol Effect on Arterial Oxygenation in COPD Patients During One-lung Ventilation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4-2023-0242
Record Dates: First submitted 2023-06-13; First posted 2023-06-22 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: One-lung Ventilation; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Normal saline
  Interventions: Drug: 5ml of inhaled normal saline
- Salbutamol group (Experimental): Salbutamol + normal saline
  Interventions: Drug: 2.5mg (2.5ml) of inhaled salbutamol and 2.5ml of inhaled normal saline

INTERVENTIONS:
Drug: 5ml of inhaled normal saline — After the initiation of OLV, 5ml of normal saline is inhaled for 20 minutes using ultrasonic nebulizer, which is connected to the inspiratory limb of the ventilator system. Arterial blood gas analysis is performed 30 minutes after the completion of drug inhalation.
  Arms: Control group
Drug: 2.5mg (2.5ml) of inhaled salbutamol and 2.5ml of inhaled normal saline — After the initiation of OLV, mixture of salbutamol 2.5mg and normal saline 2.5ml is inhaled for 20 minutes using ultrasonic nebulizer, which is connected to the inspiratory limb of the ventilator system. Arterial blood gas analysis is performed 30 minutes after the completion of drug inhalation.
  Arms: Salbutamol group

SUMMARY:
One-lung ventilation (OLV) is essential part of anesthesia during thoracic procedures. However, OLV induces a drastic increase of intrapulmonary shunt due to maintained pulmonary perfusion through the nonventilated lung, which may result in severe hypoxemia. Although the protective mechanisms of hypoxic pulmonary vasoconstriction favorably modulate pulmonary perfusion to the ventilated lung, the effect is attenuated in patients with history of chronic obstructive pulmonary disease (COPD), which alters compliance of the pulmonary artery.

Salbutamol is a selective short-acting beta2-agonist and when inhaled during OLV, it acts selectively on the pulmonary vasculature reducing pulmonary vascular resistance of well-ventilated lung. We hypothesized that inhaled salbutamol would alleviate ventilation-perfusion mismatch during OLV of COPD patients, and aimed to assess the effects of salbutamol on oxygenation in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 40~80yrs, scheduled for videoscope-assisted pulmonary lobectomy
* American Society of Anesthesiologists Class III 또는 IV
* Moderate or more severe COPD according to GOLD criteria (FEV1/FVC<70%, FEV1<80%)

Exclusion Criteria:

* New York Heart Association class >II
* AST level ≥100 IU/mL or ALT ≥ level 50 IU/L
* Creatinine clearance < 30mL/min
* History of severe coronary artery occlusive disease, unstable angina, or recent myocardial infarction within 6 months
* History of pulmonary hypertension or pulmonary edema
* History of cerebrovascular accident within 3 months

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-07-21 (Estimated)

PRIMARY OUTCOMES:
PaO2 (partial pressure of arterial oxygen) to FiO2 (fraction of inspired oxygen) ratio (P/F ratio) | Thirty minutes after the completion of drug inhalation
  The P/F ratio is a widely-used objective tool to identify hypoxemic respiratory failure when supplemental oxygen has been administered. It can be used to evaluate the effect of salbutamol on oxygenation during OLV.

CONTACTS AND LOCATIONS:
Overall Officials: Young Jun Oh, Principal Investigator — Department of Anesthesiology and Pain Medicine, Severance Hospital, Yonsei University Health System, Seoul, Korea
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No